CLINICAL TRIAL: NCT06431113
Title: Effect of Fixed Combination Citicoline 500 mg, Homotaurine 50 mg, Pyrroloquinoline Quinone (Neuprozin Mito®) on Pattern Electroretinogram in Controlled Open Angle Glaucoma Patients:A Multicenter, Randomized, Single Blind, Cross-over Study
Brief Title: Effect of Fixed Combination Citicoline Homotaurine and Pyrroloquinoline Quinone on Pattern-electroretinogram in Glaucoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Collaborators: Federico II University (Other); University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Gemma Caterina Maria Rossi, Principal investigator, Ophthalmologist, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NP-MITO
Record Dates: First submitted 2024-05-21; First posted 2024-05-28 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2024-05

CONDITIONS: Glaucoma; Neuroprotection
Keywords: glaucoma; neuroprotection; citicoline; homotaurine; Pyrroloquinoline quinone; visual field; pattern electroretinogram; oct; quality of life
MeSH Terms: conditions — Glaucoma; Ornithine Carbamoyltransferase Deficiency Disease | interventions — Cytidine Diphosphate Choline; tramiprosate; PQQ Cofactor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Citicoline 500 mg+Homotaurine 50 mg+Pyrroloquinoline quinone (Neuprozin Mito®-NPM) (Experimental): Citicoline 500 mg plus Homotaurine 50 mg plus Pyrroloquinoline quinone (Neuprozin Mito® - NPM) fixed combination for 4 months followed by Cebrolux -CIT for 4 months, besides standard topical treatment
  Interventions: Combination Product: Citicoline 500 mg plus Homotaurine 50 mg plus Pyrroloquinoline quinone (Neuprozin Mito® )
- Cebrolux -CIT for 4 months (Active Comparator): Citicoline 800 (Cebrolux-CIT) for 4 months followed by Citicoline 500 mg plus Homotaurine 50 mg plus Pyrroloquinoline quinone (Neuprozin Mito® - NPM) for 4 months, besides standard topical treatment
  Interventions: Combination Product: Citicoline 500 mg plus Homotaurine 50 mg plus Pyrroloquinoline quinone (Neuprozin Mito® )

INTERVENTIONS:
Combination Product: Citicoline 500 mg plus Homotaurine 50 mg plus Pyrroloquinoline quinone (Neuprozin Mito® ) — treatment for 4 months and then cross over to the other therapy

SUMMARY:
The goal of this clinical trial is to examine the effect of the fixed combination Citicoline 500 mg, Homotaurine 50 mg, Pyrroloquinoline quinone (PQQ) disodium salt (Neuprozin Mito®) on pattern electroretinogram (PERG) in patients with primary open angle glaucoma on well controlled intraocular pressure It will also learn about the safety of this fixed combination. The main questions it aims to answer are:

Does the fixed combination Citicoline 500 mg, Homotaurine 50 mg, Pyrroloquinoline quinone (PQQ) disodium salt (Neuprozin Mito®) improve PERG amplitude and/or latency? Does the fixed combination act as neuromodulator in glaucoma patients based on electrophysiology? Does the fixed combination improve quality of life of glaucoma patients? Does the fixed combination have any effect on optical coherence tomography (OCT)?

Researchers will compare the fixed combination Citicoline 500 mg, Homotaurine 50 mg, Pyrroloquinoline quinone (PQQ) disodium salt (Neuprozin Mito®) to citicoline 800 mg to see if the fixed combination works better than citicoline alone as neuroprotective agent in glaucoma.

Participants will:

Take the fixed combination or citicoline alone every day for 4 months After 4 months patients will be crossed over to the other treatment for 4 months.

Visit the clinic at enrollment and once every 4 months (at month 4 and at month 8) for checkups and tests (visual field, OCT, PERG and quality of life questionnaire)

DETAILED DESCRIPTION:
Our general purpose is to evaluate the potential beneficial effects of supplementation of a fixed combination of Citicoline 500 mg plus Homotaurine 50 mg plus Pyrroloquinoline quinone on retinal ganglion cells (RGCs) function in subjects with glaucoma by pattern electroretinogram.

Primary objective To compare the effects of adding the fixed combination of Citicoline 500 mg plus Homotaurine 50 mg plus Pyrroloquinoline quinone (Neuprozin Mito® - NPM) a tablet a day on PERG examination (p50 wave) at four months of therapy, compared to citicoline 800 mg alone (Cebrolux® - CIT), as add-on to standard topical therapy.

Secondary objectives

To compare the two treatments (Neuprozin Mito® - NPM vs citicoline - CIT - alone) in terms of:

* visual acuity over time
* visual field changes over time, if any
* Quality of Life perception (National Eye Institute-Visual function questionnaire 25 item -NEI VFQ25 questionnaire) over time
* optical coherence tomography - OCT- changes over time, if any

  * Safety (Incidence of adverse events)

Study design and planning Multicentric, randomized, 2-sequence, 2-period, 2-treatment, crossover study, with blind outcome assessor.

Centers

1. Azienda Ospedaliera Universitaria Federico II ; UOC Oculistica, Napoli
2. Clinica Oculistica dell'Università degli Studi di Pavia, IRCCS Policlinico San Matteo Foundation, Pavia.
3. Dipartimento di Scienze Medico-Chirurgiche e Medicina Traslazionale, Università di Roma "Sapienza", Roma

Study duration Study duration ; 14 months Enrolment period: 6 months Minimum Follow-up: 8 months Total sample size: 40 patients

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years;
* diagnosis of primary OAG (POAG) from, at least, 3 years;
* visual acuity > 0.7 (7/10) decimals;
* refractive error < 5 Diopter (D) (spheric) and < 2D (toric);
* transparent diopter means (cornea and lens);
* controlled intraocular pressure (IOP) (<18 mmHg, morning value) with prostaglandin analogues as monotherapy;
* stable intraocular pressure - IOP < 18 mmHg in the last 2 years;
* stable and unchanged topical therapy in the last 6 months;
* at least two reliable visual fields (Humphrey 24-2 Swedish interactive threshold algorithm-SITA Standard) per year in the last 2 years;
* early to moderate visual field defect (mean deviation, MD <12 dB);
* electrophysiological (pattern electroretinogram-PERG) parameters alterations similar to glaucomatous pathology;
* written consent to participate to study procedures and data utilization in an anonymous form

Exclusion Criteria:

* ocular hypertension with normal optic nerve and visual field; angle closure glaucoma; congenital glaucoma; secondary glaucoma; normal tension glaucoma;
* history of recurrent uveitis/scleritis/herpes infection;
* pregnancy and breastfeeding;
* contraindication to Citicoline and/or Homotaurine and/or pyrroloquinoline quinone -PQQ
* contraindication to prostaglandine analogues
* topical therapy with Brimonidine or beta-blockers as monotherapy or fixed combination
* topical therapy with pilocarpine and aceclidine, monotherapy or fixed combination
* systemic or topical treatment with another neuroprotective agent in the last 4 months prior to enrollment
* systemic betablockers
* systemic therapies affecting patients' performance in visual field examination (sedatives);
* glaucomatous scotomas within 10 degree from fixation
* any condition limiting the patient's ability to participate in the study;
* other ocular causes of visual field and PERG changes, such as cataract, myopic chorioretinopathy, macular diseases, retinal vascular occlusion, diabetic retinopathy;
* other systemic causes of visual field and PERG changes such as neurodegenerative disorders (Alzheimer's disease, Parkinson's disease, acute lateral sclerosis, multiple sclerosis) or pituitary disorders;
* cerebral ischemia in the last 2 years
* any change in topical therapy in the 6 months prior to enrollment or during the study period
* concomitant participation to another clinical trial
* any previous filtering and/or retinal surgery;
* cataract surgery in the last 6 months;
* any previous laser treatment for glaucoma in the last 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-01-27 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
To compare the effects of adding the fixed combination of Citicoline 500 mg+Homotaurine 50 mg+Pyrroloquinoline quinone (Neuprozin Mito® - NPM) on pattern-electroretinogram -PERG- amplitudes | 4 months
  amplitude of PERG waves (microVolt)
To compare the effects of adding the fixed combination of Citicoline 500 mg+Homotaurine 50 mg+Pyrroloquinoline quinone (Neuprozin Mito® - NPM) on PERG latencies | 4 months
  latency of PERG waves (milliseconds)

SECONDARY OUTCOMES:
To compare the two treatments in terms of: • visual acuity over time | 4 months
  visual acuity evaluation
To compare the two treatments in terms of: • visual field changes over time, if any | 4 months
  Pattern Standard Deviation and Mean Deviation (deciBell)
To compare the two treatments in terms of: • Quality of Life perception national eye institute-visual function questionnaire 25 items (NEI VFQ25) over time | 4 months
  quality of life with questionnaire national eye institute-visual function questionnaire 25 items (NEI-VFQ25) (from 0=worst score/quality of life to 100 better score/quality of life)
To compare the two treatments in terms of: • optical coherence tomography - OCT changes over time, if any | 4 months
  retinal nerve fiber layer (RNFL) and ganglion cells complex (GCC)
To compare the two treatments in terms of: • Safety (Incidence of adverse events) | 8 months
  adverse events onset

CONTACTS AND LOCATIONS:
Overall Officials: Ciro Costagliola, MD, Principal Investigator — Federico II University eye Clinic, Naples
Locations (2):
- Italy (2):
  - Clinica Oculistica Università Federico II, Napoli, Napoli
  - Gemma Caterina Maria Rossi, Pavia, PV